CLINICAL TRIAL: NCT06466967
Title: Clinical Utility of a Tight Glucose Objectives Through Advanced Hybrid Closed-loop Systems in Adult Patients With Type 1 Diabetes and Poor Glycemic Control
Brief Title: Clinical Utility of Tight Objectives of Advanced Hybrid Closed-loop Systems Among Type 1 Diabetes Patients (TightT1AHCL)
Acronym: TightT1AHCL
Status: Recruiting | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: CI-712
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; advanced hybrid closed-loop; tight time in range; artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Type 1 diabetes patients treated with AHCL (CamAPS-Ypsopump): Patients with type 1 diabetes on treatment with AHCL (CamAPS-Ypsopump) and a strict programmed glucose target (80-99 mg/dL).
  Interventions: Device: Advanced hybrid closed-loop CamAPS FX

INTERVENTIONS:
Device: Advanced hybrid closed-loop CamAPS FX — Treatment with a strict programmed glucose target (80-99 mg/dL).
  Other Names: Ypsopump; CamAPS FX

SUMMARY:
Diabetes is a chronic disease with a relevant public health burden. Maintaining blood glucose levels as close to normal as possible is essential to avoid the associated microvascular and macrovascular complications. Therefore, the key to prevent and/or reduce the development of these chronic complications lies in an adequate and strict glycemic control.

This study consist of a prospective analytical clinical study in patients with type 1 diabetes (T1D). The main objective is to analyze the effect on time in range (TIR, 70-180 mg/dL) of interstitial glucose after switching to a tighter glucose objective in advanced hybrid closed-loop (AHCL) treated adult T1D patients previously treated with multiple dose insulin injection (MDI) or other AHCL systems without tighter glucose objective function.

DETAILED DESCRIPTION:
Diabetes is a chronic disease with a relevant public health burden. T1D is characterized by the autoimmune destruction of insulin-producing pancreatic beta cells, which requires the administration of exogenous insulin for its treatment. Maintaining blood glucose levels as close to normal as possible is essential to avoid the associated microvascular and macrovascular complications that affect quality of life, as well as morbidity and mortality due to the deleterious long-term effects of suboptimal control. Therefore, the key to prevent and/or reduce the development of these complications lies in adequate and strict glycemic control.

On the one hand, the use of advanced hybrid closed-loop (AHCL) systems in patients with T1D is associated with improved glycemic control and quality of life in both controlled clinical trials and real-life studies. Since 2021, AHCL systems are considered the standard of care, ahead of traditional MDI. On the other hand, among the adjustment parameters of these systems, each AHCL offers different target levels of glycemic control. There is previous evidence that correlates the use of the more intense modes offered by each of the systems with substantial increases in TIR, improvement in the other glycometric variables, as well as the development of acute or chronic complications. In this regard, a new AHCL system has recently been introduced in Spain: CamAPS FX. It is the first AHCL system with the availability of setting lycemic control targets below the traditional 100 mg/dL limit. This system allows glycemic objective as low as 80 mg/dL.

However, there is no information on the benefits and safety of using tighter control targets. The main objective of this study is to analyze the effect on TIR after switching to a tighter glucose objective throught AHCL among adult T1D patients previously treated with MDI or other AHCL systems without this feature.

This is monocenter prospective analytical clinical study (non-randomized). The target population will be adult T1D patients not meeting glycemic control goals followed in Ciudad Real General University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes.
* Age greater than or equal to 18 years.
* HbA1c > 7% (previous poor glycemic control condition).
* Prior treatment with MDI or aHCL.

Exclusion Criteria:

* Other types of diabetes.
* Pregnancy or pre-conception control.
* Uncontrolled psychiatric disease.
* Current or previous treatment with CamAPS-Ypsopump.
* No glucometric data available during the periods under study.
* History of severe hypoglycemia.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 1 diabetes and poor prior glycemic control, regardless previous treatment, attended in the Public Health System of Castilla-La Mancha in the Health Area of the Ciudad Real General University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Time in Range (TIR) differences | 3 months
  Percentage differences in time in range (TIR, 70-180 mg/dL) of interstitial glucose after switching to AHCL with tighter glycemic control targets.

SECONDARY OUTCOMES:
Time in Range (TIR) differencies among therapies | 3 months
  Percentage differences in time in range (TIR 70-180 mg/dL) of interstitial glucose after switching to AHCL with tighter glycemic control targets depending on previous therapy: multi-dose insulin or other AHCL systems with less stringent objectives.
Differences between stringent glucose control targets | 3 months
  To analyze the possible differences on time in range (TIR) using different interstitial glucose targets (from 80 to 99 mg/dL).
HbA1c differences | 3 months
  Differences in HbA1c values after switching to AHCL with tighter glycemic control targets.
Usage of AHCL system | 3 months
  To assess the effect on the time spent using AHCL systems after switching: percentage of time spent using the AHCL system.
MCG adherence | 3 months
  To assess the effect on the time of use of MCG after switching: percentage of MCG sensor activity time.
Total daily insulin requirements | 3 months
  To assess the effect on total daily insulin requirements after switching to AHCL therapy with tighter glycemic objective.
Basal daily insulin requirements | 3 months
  To assess the effect on basal insulin requirements after switching to AHCL therapy with tighter glycemic objective.
Bolus daily insulin requirements | 3 months
  To assess the effect on insulin bolus requirements after switching to AHCL therapy with tighter glycemic objective.
Time in Tight Range (TTIR 70-140 mg/dL) differences | 3 months
  Percentage differences in time in tight range (TIR 70-140 mg/dL) of interstitial glucose after switching to AHCL with stringent glycemic control targets.
Time Above Range 1 (TAR-1 >180 mg/dL) differences | 3 months
  Percentage differences in Time Above Range 1 (TAR-1 >180 mg/dL) of interstitial glucose after switching to AHCL with stringent glycemic control targets.
Time Above Range 2 (TAR-2 >250 mg/dL) differences | 3 months
  Percentage differences in Time Above Range 2 (TAR-2 >250 mg/dL) of interstitial glucose after switching to AHCL with stringent glycemic control targets.
Time Below Range 1 (TBR-1 <70 mg/dL) differences | 3 months
  Time and percentage differences in Time Below Range 1 (TBR-1 <70 mg/dL) of interstitial glucose after switching to AHCL with stringent glycemic control targets.
Time Below Range 2 (TBR-2 <54 mg/dL) differences | 3 months
  Time and percentage differences in Time Below Range 2 (TBR-2 <54 mg/dL) of interstitial glucose after switching to AHCL with stringent glycemic control targets.
Episodes of hyperglycemia level 1 (nº of episodes >180 mg/dL). | 3 months
  Episodes of hyperglycemia level 1 (nº of episodes >180 mg/dL) after switching to aHCL with stringent glycemic control targets.
Episodes of hyperglycemia level 2 (nº of episodes >250 mg/dL). | 3 months
  Episodes of hyperglycemia level 2 (nº of episodes >250 mg/dL) after switching to AHCL with stringent glycemic control targets.
Episodes of hypoglycemia level 1 (nº of episodes <70 mg/dL). | 3 months
  Episodes of hypoglycemia level 1 (nº of episodes <70 mg/dL) after switching to AHCL with stringent glycemic control targets.
Episodes of hypoglycemia level 2 (nº of episodes <54 mg/dL). | 3 months
  Episodes of hypoglycemia level 2 (nº of episodes <54 mg/dL) after switching to AHCL with stringent glycemic control targets.
Nocturnal episodes of hypoglycemia | 3 months
  Nocturnal episodes of hypoglycemia (nº of episodes <70 and <54 mg/dL) after switching to AHCL with stringent glycemic control targets.
Glycemic variability | 3 months
  Glycemic variability (measured throught percentage of the coefficient of variation, CV) differences after switching to AHCL with stringent glycemic control targets.
Mean interstitial glucose | 3 months
  Mean interstitial glucose differences after switching to AHCL with stringent glycemic control targets.
Glucose management indicator (GMI) | 3 months
  Glucose management indicator (GMI) differences after switching to AHCL with stringent glycemic control targets.
Acute complications and mortality | 3 months
  Analyzing the impact of the switch on the frequency of acute complications and mortality due to T1D: severe hypoglycemia, non-acidotic ketotic hyperglycemia, diabetic ketoacidosis, hospital admissions and deaths.
Differences in the Percetage of patients fullfilling the International Consensus of Time in Range | 3 months
  Differences in the Percetage of patients fullfilling the International Consensus of Time in Range (TAR2 <5%, TAR1 <25%, TIR >70%, TBR1 <4%, TBR2 <1%, CV>36%).

OTHER OUTCOMES:
Hypoglycemia Fear Survey (HFS questionnaire) | 3 months
  Assessing the fear of hypoglycemia according to the HFS questionnaire (with values between 24 points and a maximum of 120 indicating a high fear of hypoglycemia) after switching to AHCL with stringent glycemic control targets.
Diabetes Treatment Satisfaction Questionnaire (DTSQ) | 3 months
  Assessing the satisfaction with treatment according to the DTSQ questionnaire (options graduated from 0 to 6 from the lowest to the highest degree of satisfaction, with a minimum of 0 and a maximum of 12) after switching to AHCL with stringent glycemic control targets.
Clarke's questionnaire | 3 months
  Assessing the awareness of hypoglycemia according to Clarke's questionnaire (indicates high risk of inadvertent hypoglycemia with a score equal to or greater than four) afterswitching to AHCL with stringent glycemic control targets.
Quality-of-life questionnaire designed for diabetes mellitus (EsDQOL) | 3 months
  Assessing the perceived quality of life according to the EsDQOL questionnaire (with values between 46 and a maximum of 230 which would indicate poor satisfaction with current treatment) after switching to AHCL with stringent glycemic control targets.

CONTACTS AND LOCATIONS:
Locations (1):
- Ciudad Real General University Hospital, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Undecided
According to the requested data.

REFERENCES:
- [Background] Battelino T, Danne T, Bergenstal RM, Amiel SA, Beck R, Biester T, Bosi E, Buckingham BA, Cefalu WT, Close KL, Cobelli C, Dassau E, DeVries JH, Donaghue KC, Dovc K, Doyle FJ 3rd, Garg S, Grunberger G, Heller S, Heinemann L, Hirsch IB, Hovorka R, Jia W, Kordonouri O, Kovatchev B, Kowalski A, Laffel L, Levine B, Mayorov A, Mathieu C, Murphy HR, Nimri R, Norgaard K, Parkin CG, Renard E, Rodbard D, Saboo B, Schatz D, Stoner K, Urakami T, Weinzimer SA, Phillip M. Clinical Targets for Continuous Glucose Monitoring Data Interpretation: Recommendations From the International Consensus on Time in Range. Diabetes Care. 2019 Aug;42(8):1593-1603. doi: 10.2337/dci19-0028. Epub 2019 Jun 8. PMID 31177185
- [Background] Bally L, Thabit H, Kojzar H, Mader JK, Qerimi-Hyseni J, Hartnell S, Tauschmann M, Allen JM, Wilinska ME, Pieber TR, Evans ML, Hovorka R. Day-and-night glycaemic control with closed-loop insulin delivery versus conventional insulin pump therapy in free-living adults with well controlled type 1 diabetes: an open-label, randomised, crossover study. Lancet Diabetes Endocrinol. 2017 Apr;5(4):261-270. doi: 10.1016/S2213-8587(17)30001-3. Epub 2017 Jan 14. PMID 28094136
- [Background] Brown SA, Kovatchev BP, Raghinaru D, Lum JW, Buckingham BA, Kudva YC, Laffel LM, Levy CJ, Pinsker JE, Wadwa RP, Dassau E, Doyle FJ 3rd, Anderson SM, Church MM, Dadlani V, Ekhlaspour L, Forlenza GP, Isganaitis E, Lam DW, Kollman C, Beck RW; iDCL Trial Research Group. Six-Month Randomized, Multicenter Trial of Closed-Loop Control in Type 1 Diabetes. N Engl J Med. 2019 Oct 31;381(18):1707-1717. doi: 10.1056/NEJMoa1907863. Epub 2019 Oct 16. PMID 31618560
- [Background] Bergenstal RM, Nimri R, Beck RW, Criego A, Laffel L, Schatz D, Battelino T, Danne T, Weinzimer SA, Sibayan J, Johnson ML, Bailey RJ, Calhoun P, Carlson A, Isganaitis E, Bello R, Albanese-O'Neill A, Dovc K, Biester T, Weyman K, Hood K, Phillip M; FLAIR Study Group. A comparison of two hybrid closed-loop systems in adolescents and young adults with type 1 diabetes (FLAIR): a multicentre, randomised, crossover trial. Lancet. 2021 Jan 16;397(10270):208-219. doi: 10.1016/S0140-6736(20)32514-9. PMID 33453783
- [Background] Beato-Vibora PI, Chico A, Moreno-Fernandez J, Bellido-Castaneda V, Nattero-Chavez L, Picon-Cesar MJ, Martinez-Brocca MA, Gimenez-Alvarez M, Aguilera-Hurtado E, Climent-Biescas E, Azriel-Mir S, Rebollo-Roman A, Yoldi-Vergara C, Pazos-Couselo M, Alonso-Carril N, Quiros C. A Multicenter Prospective Evaluation of the Benefits of Two Advanced Hybrid Closed-Loop Systems in Glucose Control and Patient-Reported Outcomes in a Real-world Setting. Diabetes Care. 2024 Feb 1;47(2):216-224. doi: 10.2337/dc23-1355. PMID 37948469
- [Background] El Malahi A, Van Elsen M, Charleer S, Dirinck E, Ledeganck K, Keymeulen B, Crenier L, Radermecker R, Taes Y, Vercammen C, Nobels F, Mathieu C, Gillard P, De Block C. Relationship Between Time in Range, Glycemic Variability, HbA1c, and Complications in Adults With Type 1 Diabetes Mellitus. J Clin Endocrinol Metab. 2022 Jan 18;107(2):e570-e581. doi: 10.1210/clinem/dgab688. PMID 34534297